CLINICAL TRIAL: NCT05087095
Title: Managing Distress in Malignant Brain Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-21-18040
Record Dates: First submitted 2021-08-26; First posted 2021-10-21 (Actual); Results first posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Cancer Metastatic to Brain; Brain Metastases, Adult
Keywords: bMET; CALM; Service Members; Veterans
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CALM (Experimental): CALM therapy will be provided via telehealth. Participants will complete surveys (post-session, post-intervention, and 90-day follow-up) via secure email link. Exit interviews will be conducted by phone
  Interventions: Behavioral: CALM Intervention

INTERVENTIONS:
Behavioral: CALM Intervention — The CALM intervention includes 6 individual therapy sessions, each approximately 45-60 minutes in length, delivered over 3 months. Participants will be asked to complete self-report surveys of behavioral and psychological variables surveys at the following timepoints:
  * Within one week before initiating the CALM intervention therapy
  * Within one week after its completion,
  * 3 months after the CALM intervention is complete
    * After each intervention session, participants will complete a brief post-session survey to assess acceptability of CALM session components

SUMMARY:
To identify potential adaptations of the managing cancer and living meaningfully (CALM) intervention that will be required for service members, Veterans, their beneficiaries, and civilian cancer metastasis to the brain (bMET) populations.

DETAILED DESCRIPTION:
Single-arm, mixed-methods, Phase IIa, proof-of-concept trial to inform CALM adaptations for service members (SMs), Veterans, their beneficiaries, and civilians with bMET.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of brain metastasis (bMET) confirmed via medical records, radiography or histopathology
* At least 2 weeks post-surgical cranial resection or cranial biopsy (if applicable)
* Score > 20 on the TICS
* Report elevated depression (PHQ-9 score ≥ 10) OR death anxiety symptoms (DADDS score ≥ 15)
* Ability to read, speak, and understand English
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Major communication difficulties, which would prohibit psychotherapeutic interaction
* Inability to meet with interventionist via an electronic device for telehealth intervention sessions
* Inability to understand and provide informed consent
* Medical, psychological, or social condition that, in the opinion of the investigator, may increase the participant's risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashlee Loughan, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) to other researchers at this time.

REFERENCES:
- [Derived] Loughan AR, Lanoye A, Willis K, Braun SE, Davies A, Rodin G, Thacker L, Fox A, Kleva C, Zarrella G, Mazzeo S, Svikis D, Swartz L. Managing Cancer and Living Meaningfully in adults with brain metastases: A NIH ORBIT model phase II feasibility and proof-of-concept trial. Neurooncol Pract. 2024 Oct 15;12(2):271-280. doi: 10.1093/nop/npae097. eCollection 2025 Apr. PMID 40110068

RESULTS

PARTICIPANT FLOW:
Groups:
- CALM: CALM therapy will be provided via telehealth. Participants will complete surveys (post-session, post-intervention, and 90-day follow-up) via secure email link. Exit interviews will be conducted by phone
  CALM Intervention: The CALM intervention includes 6 individual therapy sessions, each approximately 45-60 minutes in length, delivered over 3 months. Participants will be asked to complete self-report surveys of behavioral and psychological variables surveys at the following timepoints:
  * Within one week before initiating the CALM intervention therapy
  * Within one week after its completion,
  * 3 months after the CALM intervention is complete
    * After each intervention session, participants will complete a brief post-session survey to assess acceptability of CALM session components
Period: Overall Study
Arm/Group | CALM
Started | 13
Completed | 9
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | CALM
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants] — Population: Two participants declined to provide DOB
  Participants
    number analyzed (Participants) | 11
    <=18 years | 0
    Between 18 and 65 years | 6
    >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 10
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Assess the Need for Adaptations to the CALM Intervention as Measured by the Applicability of the 4 CALM Domains
Description: At the exit interview, participants will be asked to rate the applicability of the four CALM domains on a Likert Scale from 1 (not applicable) to 5 (very applicable). The four CALM domains are as follows: Domain 1) represents symptom management and communication with healthcare providers, Domain 2) reflects changes in personal relationships, Domain 3) sense of meaning and purpose, and Domain 4) the future, hope and mortality. Higher scores mean greater applicability.
Time Frame: 4 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CALM
Number analyzed (Participants) | 9
score on a scale
  Domain 1 | 3.2 (1.2)
  Domain 2 | 4.0 (1.3)
  Domain 3 | 4.0 (1.7)
  Domain 4 | 3.5 (1.3)

2. Primary Outcome: Feasibility of CALM Intervention in the Proof of Concept Project as Measured by the Rates of Participant Screening, Eligibility, and Consent.
Description: Determine how many patients consent to screening after referral to the program, how many patients are eligible for the program after being screened, and how many consent/enroll in the program if eligible.
Time Frame: 12 months
Population: The number of participants interested / referred for the protocol = 32. The number screened = 21
Measure: Count of Participants; unit: Participants
Arm/Group | CALM
Number analyzed (Participants) | 32
Participants
  Screened | 21
  Eligible | 13
  Consented | 13

3. Primary Outcome: Feasibility of CALM Intervention in the Proof of Concept Project as Measured by Attendance at CALM Sessions
Description: Percent of sessions attended across all participants
Time Frame: 3 Months
Measure: Number; unit: percentage of CALM sessions attended
Units Other Than Participants: Number of CALM sessions
Arm/Group | CALM
Number analyzed (Participants) | 13
Number analyzed (Number of CALM sessions) | 78
percentage of CALM sessions attended | 76

4. Primary Outcome: Feasibility of CALM Intervention in the Proof of Concept Project as Measured by the Rates of Post-session Assessment Completion
Description: Percent of post-session surveys completed by participants immediately after the intervention
Time Frame: 3 Months
Measure: Number; unit: percentage of assessments completed
Units Other Than Participants: Post-session surveys
Arm/Group | CALM
Number analyzed (Participants) | 11
Number analyzed (Post-session surveys) | 66
percentage of assessments completed | 70

5. Primary Outcome: Feasibility of CALM Intervention in the Proof of Concept Project as Measured by Post-intervention Assessment Completion
Description: Percent of post-intervention surveys completed
Time Frame: 3 Months
Measure: Number; unit: percentage of assessments completed
Arm/Group | CALM
Number analyzed (Participants) | 11
percentage of assessments completed | 82

6. Primary Outcome: Benefit of Intervention in the Proof of Concept Project
Description: Benefit will be assessed by participant responses to a question during the exit interview (e.g., Rate your overall benefit on a scale of 1-5).
Time Frame: 4 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CALM
Number analyzed (Participants) | 9
units on a scale | 4.4 (0.53)

ADVERSE EVENTS:
Time Frame: Baseline to three months
Arm/Group | CALM
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-07): https://cdn.clinicaltrials.gov/large-docs/95/NCT05087095/Prot_SAP_001.pdf
  • Informed Consent Form (2022-01-07): https://cdn.clinicaltrials.gov/large-docs/95/NCT05087095/ICF_000.pdf